CLINICAL TRIAL: NCT00662662
Title: Sexual Behavior in Head and Neck Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2007-0485
Record Dates: First submitted 2008-04-17; First posted 2008-04-21 (Estimated); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Oropharyngeal Cancer; Head and Neck Cancer; Squamous Cell Carcinoma
Keywords: Oropharyngeal Cancer; Non-Oropharyngeal Cancer; Head and Neck Cancer; Squamous Cell Carcinoma; Squamous cell carcinoma of the head and neck; SCCHN; HPV-16; Questionnaire; Sexual Behavior; Survey
MeSH Terms: conditions — Oropharyngeal Neoplasms; Head and Neck Neoplasms; Carcinoma, Squamous Cell; Squamous Cell Carcinoma of Head and Neck; Sexual Behavior | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Oropharyngeal Cancer
  Interventions: Behavioral: Questionnaire
- Non-Oropharyngeal Cancer
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — The questionnaire contains 18 questions and is estimated to take approximately 10-15 minutes to complete.

SUMMARY:
The goal of this behavioral research study is to learn if certain sexual behaviors increase the risk for developing head and neck cancers associated with a virus called human papillomavirus (HPV-16). Knowing this information could help doctors better teach patients about avoiding certain risk factors, which may help to prevent the disease.

DETAILED DESCRIPTION:
SCCHN is believed to be caused by different types of viruses being exposed to the mucous membrane on the inside of the mouth, throat, and voice box, over a long period of time. This exposure results in changes in the cells of the mouth, throat, and voice box, which can lead to the development of cancer.

HPV-16 has been linked to SCCHN. Half of all cancers of the oropharynx (the middle part of the throat, the base of the tongue, and tonsils) may be caused by HPV-16. HPV-16 is normally spread sexually, and is one of the main causes of cervical cancer in women. By finding out if the virus is also spread sexually to the throat, doctors may be able to teach patients about risk factors for developing cancer in this area.

Study Procedures:

If you agree to take part in this study, you will be asked to complete a questionnaire about your sexual history, such as specific sexual practices, number of partners, exposure to HPV and other viruses, and any medical history related to HPV-16. The questionnaire will take 10-15 minutes to complete.

None of your personal identifying information will be attached to your questionnaire, and the questionnaire will be assigned a one-of-a-kind study code number.

To check your cancer diagnosis, your medical records will be reviewed.

Length of Study:

Once you have completed the questionnaire, your participation in this study is over.

This is an investigational study.

Up to 1,500 patients will be enrolled in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with newly diagnosed, previously untreated squamous cell carcinoma of the head and neck (SCCHN) who are candidates for the molecular epidemiology study LAB00-062 of head and neck cancer.
2. Must have the ability to understand and provide informed consent.
3. Patients must be 18 years and older.
4. Ability to read, write, and speak English.
5. Resident of the United States.
6. Agrees to have tumor tissue, if available, tested for HPV. No additional biopsy will be requested.

Exclusion Criteria:

1. Previous cancer diagnosis excluding non-melanoma skin cancer.
2. Blood transfusion within the previous 6 months.
3. Immune suppression, such as HIV disease or immune-suppressing therapy (i.e., steroids).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 600 oropharynx study participants and 900 non-oropharynx study participants.
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2008-04 (Actual); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
To find out if certain sexual behaviors increase the risk for developing head and neck cancers associated with a virus called human papillomavirus (HPV-16). | 6 Years

CONTACTS AND LOCATIONS:
Overall Officials: Erich Sturgis, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org